CLINICAL TRIAL: NCT04789187
Title: Randomized Controlled Trial of Simultaneous Exercise During Neo-/Adjuvant Chemotherapy in Breast Cancer Patients and Its Effects on Neurocognition
Brief Title: Exercise, Cancer and Cognition: The ECCO-Study
Acronym: ECCO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Johannes Kepler University of Linz (Other)
Collaborators: German Sport University, Cologne (Other); University of Graz (Other); Charite University, Berlin, Germany (Other); Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Milan Vosko, MD, PhD, Principal Investigator, Johannes Kepler University of Linz
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1191/2018
Record Dates: First submitted 2020-03-08; First posted 2021-03-09 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Breast Cancer
Keywords: Breast; Cancer; CRCI; Chemobrain; Cognition; Exercise; High-Intensity-Interval-Training
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Chemotherapy-Related Cognitive Impairment; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Pseudonymization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Exercise intervention arm (Active Comparator)
  Interventions: Procedure: High-Intensity-Interval-Training
- Arm B: Control arm (Placebo Comparator)
  Interventions: Procedure: General Physical Activity Recommendations

INTERVENTIONS:
Procedure: High-Intensity-Interval-Training — Defined exercise program up to four times per week including high-intensity-interval-training for one year of active study intervention.
  Arms: Arm A: Exercise intervention arm
Procedure: General Physical Activity Recommendations — Patients will be given general physical activity recommendations during chemotherapy.
  Arms: Arm B: Control arm

SUMMARY:
The "ECCO"-study evaluates the efficacy of simultaneous controlled exercise during neo/-adjuvant chemotherapy in breast cancer patients and its effects on neurocognition.

In this study the investigators examine the benefits of the individualized high intensity training program on a cancer related cognitive impairment.

Changes in patients' cognition are evaluated by neuropsychological testing. Possible structural changes are detected with MRI volumetry. Biomarkers connected to Cancer Related Cognitive Impairment (CRCI) and chemotherapy related inflammatory processes which impair cognition, respectively, will be assessed.

DETAILED DESCRIPTION:
Background: Epidemiological research indicates that increased levels of physical activity are associated with decreased breast cancer risk and mortality. Thereby, exercise programs can substantially increase patients' quality of life during and after treatment. Up to 80% of breast cancer patients demonstrate a decrease in their cognitive capacity, summarized as the symptom-complex "Cancer Related Cognitive Impairment (CRCI)". Most frequently reported impairments are mild to moderate deficits in processing speed, attention, memory and executive functions. In about 35% of affected patients, cognitive symptoms persist for months, or even years, after completion of medical treatment, impairing daily functioning, limiting ability to return to work and decreasing overall quality of life. Recent studies indicate a key role of inflammatory pathways in the CRCI genesis. Attention to physical activity therefore as a potential supportive care option is increasing. Anyhow, evidence for positive effects of exercise on CRCI is still lacking.

Patients and Methods: This prospective, two-arm, 1:1 randomized, controlled trial aims to investigate the influence of high-intensity training interventions accompanying neo/-adjuvant chemotherapy on CRCI in 126 patients with early breast cancer on cognitive performance measured by the California Verbal Learning Test (CVLT). Secondary endpoints include subjective markers and tests for cognitive performance and inflammatory biomarkers as TNF-α, IL-6, IL-1α, IL-1ß which are suspected to be involved in the pathogenesis of CRCI. As cognitive impairments are believed to be connected to either functional and/or morphological hippocampal damage due to chemotherapy, head MRIs and hippocampal volume measurements will be performed. In addition to a heart rate controlled home-based endurance and strength training for one year, participants in the intervention group will perform a supervised high-intensity interval training (HIIT) exercise program at least once a week. This study will help to clarify whether a long-term supervised exercise intervention program affects CRCI in breast cancer patients and help to reason underlying mechanisms and the pathogenesis of the chemobrain.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed breast cancer and planned neo- and adjuvant chemotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Age 18 - 70 years
* Adequate hematologic functions 28d prior to randomization (Platelet count over 50 G/L, Hemoglobin over 8 g/dL)
* Able to perform exercise according to protocol
* Signed informed consent prior to randomization
* Fluid in German

Exclusion Criteria:

* Significant comorbid conditions precluding participation in a physical activity program (investigators decision)
* Anamnestic cognitive impairment or psychological disorders
* Disabled patients unable to participate in the physical activity program or performing cognitive tests
* Vigorous physical activity of >300 minutes weekly within the last year before diagnosis of breast cancer 8.3
* Patients unwilling to complete endurance exercise or complete all questionnaires related to the study
* Past or current history of other malignant neoplasms other than breast cancer in the last 5 years except basal cell carcinoma of the skin and/or in situ carcinoma of the cervix
* Clinically significant cardiovascular disease (including myocardial infarction < 6 month before randomization, unstable angina, symptomatic congestive heart failure NYHA II-IV, serious uncontrolled cardiac arrhythmia, preexcitation syndromes (eg Wolff-Parkinson-White-Syndrome), high grade or complete AV-Block, left bundle branch block, permanent pacemaker stimulation, uncontrolled hypertension (systolic blood pressure >160 mmHg), aortic valve stenosis, moderate to high-grade valve disease, endo-, myo-, pericarditis, acute aortic dissection, acute pulmonary embolism, acute phlebothrombosis of the lower extremity
* Current pregnancy or plans to become pregnant within the next year after study entry (Pregnancy tests are included in clinical routine before every chemotherapy)
* Signs of severe morphological brain damage in the baseline screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Cognition | 12 month
  The primary endpoint is measured by the changes in the total score of the California Verbal Learning Test (CVLT), measured 12 months after baseline assessment. Total points of the score are 176 pts., with less points indicating a worse outcome/ cognitive impairment and more points a better outcome/ cognitive function.

SECONDARY OUTCOMES:
Hippocampal Volume | 12 month
  Devation of hippocampal volume measured 12 months after baseline assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Milan R Vosko, MD, PhD, Study Chair — Johannes Kepler University of Linz
Locations (1):
- Kepler University Hospital, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kiesl D, Kuzdas-Sallaberger M, Fuchs D, Brunner S, Kommenda R, Tischler C, Hornich H, Akbari K, Kellermair J, Blessberger H, Ocenasek H, Hofmann P, Zimmer P, Vosko MR. Protocol for the Exercise, Cancer and Cognition - The ECCO-Study: A Randomized Controlled Trial of Simultaneous Exercise During Neo-/Adjuvant Chemotherapy in Breast Cancer Patients and Its Effects on Neurocognition. Front Neurol. 2022 Mar 25;13:777808. doi: 10.3389/fneur.2022.777808. eCollection 2022. PMID 35401389